CLINICAL TRIAL: NCT05655390
Title: Safety Intervention for Improving Functioning in Suicidal Attempters
Acronym: STRONG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB2022_0659
Record Dates: First submitted 2022-10-25; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-10

CONDITIONS: Suicide, Attempted; Functioning, Psychosocial
Keywords: suicide; cognition; neuroimaging; psychosocial functioning; quality of life
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Intervention Model Description: Experimental randomized clinical study. Rater-blinded. Sample: Suicidal attempters.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (No Intervention): (TAU)
- Intervention Group (Experimental): Treatment As Usual + Safety Intervention Planning.
  Interventions: Behavioral: Safety Intervention Planning

INTERVENTIONS:
Behavioral: Safety Intervention Planning — The therapy is based on the iFightDepression platform implemented by the European Alliance against Depression. The aim of this specific therapy is to help individuals to acquire strategies to regulate emotions and learn to tolerate discomfort preventing the imminent risk for suicidal behavior. The safety planning intervention will be conducted by identifying warning signs and provide each individual with personal and individualized coping strategies and sources of support. Main skills to be acquired and integrated for the individual are as it follows: 1) Contingency plan by five steps (identification of warning signs; applying internal coping strategies; network as distraction; safe environment; reasons for living and contact professionals), 2) Mindfulness, 3) Discomfort tolerance, and 4) Regulating emotions.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of a safety planning intervention in suicidal attempters by improving their psychosocial functional outcome and therefore enhancing their ability to perform the activities of daily living. As secondary objectives, assessment of the effectiveness of a safety planning intervention in suicidal attempters will be performed by determining cognitive performance (particularly decision-making, inhibition and attention), quality of life, clinical state and relating all these data with neuroimaging correlates. Target neuroimaging areas will be the orbitofrontal cortex and dorsal prefrontal cortex.

DETAILED DESCRIPTION:
Design: STRONG is a single-centre experimental randomized clinical trial for suicidal attempters involving a safety planning intervention and 3- to 6-months follow-ups. This study will be carried out in the Bipolar and Depressive Disorders Unit, at Hospital Clínic de Barcelona. It will be rater-blinded and will include two parallel arms (1:1) in order to assess the efficacy of a safety planning intervention compared with treatment as usual. This project has been approved by the Ethical Committee of the Hospital Clinic of Barcelona and it will be carried up in accordance with the ethical principles of the Declaration of Helsinki and Good Clinical Practice in compliance with the data protection law in force and anonymization of the collected information.

Procedures: Subsequent to signing the informed consent, a complete baseline evaluation will be carried out which includes acquisition of socio-demographic and clinical variables, psychosocial functioning, cognitive performance, quality of life assessment and neuroimaging determinations (v0). Thereafter, the whole sample will be randomized in two groups of 60 participants by parallel assignment. A group of 60 people will exclusively receive treatment as usual (non-intervention group); whereas the other group of 60 participants will receive a safety planning intervention in addition to their treatment as usual (experimental group). After two months of finishing the intervention of 4 weeks (or three months after baseline), suicidal attempters will be reassessed from a socio-demographic, clinical, psychosocial functioning, quality of life assessment as well as brief neuropsychological evaluation (v1). The neuropsychological assessment in this point will be shorter to avoid learning effect. Five months after intervention (or 6-months after baseline), a completely socio-demographic, clinical psychosocial functioning, quality of life assessment as well as neuropsychological and neuroimaging evaluation will be carried out (v2).

Assessments:

A) Socio-demographic variables: Information on gender, age, marital status, current type of cohabitation, number of offspring (if any), educational level, years of education, employment status and socioeconomic status.

B) Clinical, psychosocial functioning, quality of life evaluation: Suicidal ideation and behaviour, clinical symptomatology, in general and depressive symptoms and anxiety symptoms in particular, lifetime history of psychiatric or medical comorbidities, diagnosis, number of hospitalizations, family history of affective and psychiatric disorders, and pharmacological treatment will be collected for all subjects, premorbid adjustment, psychosocial functioning, quality of life, impulsiveness, reflective functioning and stress associated with life events will be also assessed using standardized questionnaires. Clinical variables will be assessed at baseline, two months post-intervention and at the 6-month follow-up.

C) Neuropsychological assessment: Intelligence quotient, attention, processing speed, verbal and visual memory, working memory, and executive functions will be assessed in all subjects. The extended neuropsychological battery will be administered at baseline and at 6 months. To avoid learning effects, only some of the tests evaluating attention and executive functions will be administered in the 2-month assessment post-intervention.

D) Neuroimaging assessment: Magnetic resonance imaging (MRI) will be performed at baseline, and in the 6-month follow-up. Data acquisition will be performed using a full-body MRI scanner, a Siemens Magnetom Prisma 3 Teslas. A part from structural T1, resting-state functional MRI, and diffusion-weighted imaging, two tasks related to decision making and inhibition will be carried out. Non-contrast MRI will be used. Participants will not be exposed to radiation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Having attempted suicide
* Provide written informed consent
* No claustrophobia/metallic objects/implants

Exclusion Criteria:

* Intelligence quotient below 70 and impaired functioning
* Any medical condition that could affect neuropsychological performance (such as neurological diseases) or a history of head trauma with loss of consciousness
* Participation in any structured psychological intervention within the past 6 months
* Patients who received electroconvulsive therapy within the past 6 months
* Inability to give inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Psychosocial functioning changes in Functioning Assessment Short Test (FAST). | 2 months after intervention; 5 months after intervention
  Suicidal attempters receiving a safety planning intervention will show a decrease in FAST scores, compared to those suicidal attempters receiving treatment as usual. Lower general scores on this scale indicate better psychosocial functioning.

SECONDARY OUTCOMES:
Cognitive changes in executive functions, specifically in decision-making measured by Iowa Gambling Task (IGT). | 2 months after intervention; 5 months after intervention
  Suicidal attempters receiving a safety planning intervention will experience greater improvement in cognitive performance, particularly in decision-making compared to those suicidal attempters receiving treatment as usual. A proxy of decision-making ability is extracted by means of a formula taking into account number of safe choices minus risky selections in terms of alll choices during the task. Higher scores are related to better decision-making ability.
  Normative data has been published for Spanish population and will be used to assess improvement based on the baseline visit (vs. performance 6-month follow-up).
Cognitive changes in executive functions, specifically in impulsivity measured by Stroop Test (Stroop). | 2 months after intervention; 5 months after intervention
  Suicidal attempters receiving a safety planning intervention will experience greater improvement in cognitive performance, particularly in inhibition compared to those suicidal attempters receiving treatment as usual. Inhibitory control will be assessed by measure of interference obtained through Stroop test. Higher scores here mean better inhibitory control, thus less impulsivity.
  Normative data are taken from the original version of Stroop Test and will be used to assess improvement based on the baseline visit (vs. performance 6-month follow-up).
Cognitive changes in executive functions, specifically in attention measured by Conners' Performance Test v.5 (CPT-II). | 2 months after intervention; 5 months after intervention
  Suicidal attempters receiving a safety planning intervention will experience greater improvement in cognitive performance, particularly in attention, compared to those suicidal attempters receiving treatment as usual. Measures used to assess inattention include: omissions, commissions, Hit Reaction Time (RT), Detectability (d'), Hit RT Block Change and Hit RT Inter-Stimulus Intervals (ISI) Change by means of CPT-II. All measures taken together provide an index of inattention, which is based on T-scores. In this test, higher scores reflect greater impairment.
  Normative data has been published in CPT II V.5 and will be used to assess improvement based on the baseline visit (vs. performance 6-month follow-up).
Changes in self-reported quality of life by Quality of Life 5-Dimensions scale (EuroQoL-5D). | 2 months after intervention; 5 months after intervention
  Suicidal attempters receiving a safety planning intervention will show greater improvement in quality of life compared to those suicidal attempters receiving treatment as usual taking into account baseline measures self-reported in comparison with the following visits. This scale comprises two subscales: First subscale measures quality of life using a descriptive system by dimensions (mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression). The higher the score here, the worse the quality of life. Second subscale uses a visual analog scale from 0 to 100 for self-reporting overall quality of life. Higher scores here reflect better quality of life. All items refer to the current day.
Clinical changes in suicidal behavior assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS). | 2 months after intervention; 5 months after intervention
  Suicidal attempters receiving a safety planning intervention will not show suicidal behavior measured by C-SSRS in the two follow-up visits after intervention with Safety Planning Intervention (SPI) compared to those suicidal attempters receiving treatment as usual.
Clinical changes in depressive symptomatology assessed by Patient Health Questionnaire (PHQ-9). | 2 months after intervention; 5 months after intervention
  Patient Health Questionnaire (PHQ-9) measures frequence of depressive symptoms occurrence. Lower scores show less depressive-related symptomatology. PHQ-9 scores following intervention are expected to be lower than at baseline.
Clinical changes in anxious symptomatology assessed by Generalized Anxiety Disorder (GAD-7). | 2 months after intervention; 5 months after intervention
  Generalized Anxiety Disorder (GAD-7) measures frequence of anxious symptoms occurrence. Lower scores show less anxiety-related symptomatology. GAD-7 scores following intervention are expected to be lower than at baseline.
Changes in activation of different areas of the prefrontal cortex measured by functional Magnetic Resonance Imagining (fMRI). | 5 months after intervention
  Suicidal attempters receiving a safety planning intervention will show changes in different areas of the prefrontal cortex. Changes expected include resting and activation conditions. We expect to detect more activation in prefrontal cortex (PFC) areas such as the ventrolateral PFC (including the orbitofrontal cortex), the anterior cingulate gyrus, the dorsomedial PFC and the dorsolateral PFC in patients receiving psychological intervention (in comparison with their baseline performance in task-related fMRI). Other areas such as the amygdala and medial temporal cortex will also be explored.
  Additionally, alterations in white matter connections measures by Diffusion Weighted Imaging (DWI) and Diffusion Tensor Imagining (DTI) will be assessed at baseline and will be compared with 6-months follow up imaging acquisition.
  Moreover, possible anatomical changes in prefrontal cortex areas will be also assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Iria Grande, Principal Investigator — IDIBAPS- Hospital Clinic de Barcelona
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared only under a justified request. Names and personal data will never be displayed or shared with third parties.
  The data will be collected in an information file owned by the center. The research team undertakes to preserve the privacy of patients and the confidentiality of data, in accordance with the Organic Law 3/2018, 5th December, about Personal Data Protection.
  In case of transfer of data to third parties (external promoter to the center) these will be transferred in an encrypted system, eliminating any data that could identify the patient. Only the principal investigator and her team will have access to the list of patient identification codes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When approved by the PI. For a period of 6 months at maximum.
Access Criteria: Only coded data will be transferred to third parties and to other countries, which in no case will contain information that can directly identify the participant (such as name and surname, initials, address, social security number, etc.). In the event of such a transfer, it would be for the same purpose of the study described above and guaranteeing confidentiality.

REFERENCES:
- [Derived] Roberto N, Vazquez M, Radua J, Pariente JC, Munoz-Moreno E, Laredo C, Bracco L, Fernandez T, Martin-Parra S, Martinez-Aran A, Sanchez-Moreno J, Saiz P, Ruiz-Veguilla M, Borras R, Toll A, Elices M, Brambilla P, Courtet P, Perez-Sola V, Vieta E, Grande I. Safety intervention for improving functioning in suicidal attempters (STRONG): A secondary prevention study. Study rationale and research protocol. Span J Psychiatry Ment Health. 2023 Aug 25:S2950-2853(23)00001-7. doi: 10.1016/j.sjpmh.2023.05.001. Online ahead of print. PMID 38591829